CLINICAL TRIAL: NCT05721833
Title: Effect of Noninvasive High Frequency Oscillatory Ventilation on Improving Carbon Dioxide Clearance in COPD Patients : a Clinical Crossover Trial
Brief Title: Effect of Noninvasive High Frequency Oscillatory Ventilation on Improving CO2 Clearance in COPD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jianyi Niu, Principle investigator, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIRH-202203-1
Record Dates: First submitted 2022-11-14; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COPD Exacerbation; Non-invasive Ventilation
Keywords: Noninvasive ventilation; High frequency oscillatory ventilation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Patients were randomized to receive one hour each of the two non-invasive ventilation modes before and after, and one hour of washout after receiving the first mode of ventilation before receiving the second intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-invasive high-frequency oscillatory ventilation (Experimental): Patients were titrated for relevant parameters of non-invasive ventilation the day before the trial. In the non-invasive high-frequency oscillation ventilation mode, the support pressure is consistent with the non-invasive bi-level positive pressure mode, and the high frequency airway pressure oscillation driven by the solenoid valve is added during the expiratory phase. The amplitude is about 4cmH2O, and the oscillation frequency is about 8HZ.
  Interventions: Device: Non-invasive high-frequency oscillatory
- Bilevel positive pressure ventilation (Active Comparator): Patients were titrated for relevant parameters of non-invasive ventilation the day before the trial. Noninvasive bilevel positive pressure ventilation mode pressure titration follows previous studies.
  Interventions: Device: Noninvasive Bilevel Positive Pressure Ventilation

INTERVENTIONS:
Device: Non-invasive high-frequency oscillatory — Non-invasive high-frequency oscillatory ventilation generates high-frequency pressure fluctuations in the airway caused by the opening and closing of a solenoid valve.
  Arms: non-invasive high-frequency oscillatory ventilation
Device: Noninvasive Bilevel Positive Pressure Ventilation — Noninvasive Bilevel Positive Pressure Ventilation.
  Arms: Bilevel positive pressure ventilation

SUMMARY:
High-frequency oscillatory ventilation (HFOV), as an ideal lung-protecting ventilation method, has been gradually used in neonatal critical care treatment, and is currently recommended as a rescue method for neonatal acute respiratory distress syndrome (ARDS) after failure of conventional mechanical ventilation. . Although its ability to improve oxygenation and enhance carbon dioxide (CO2) scavenging has been repeatedly demonstrated in laboratory studies, its impact on clinical outcomes in these patients remains uncertain. Non-invasive high-frequency oscillatory ventilation (nHFOV) combines the advantages of HFOV and non-invasive ventilation methods, and has become a current research hotspot in this field. It is recommended to be used to avoid intubation after conventional non-invasive ventilation therapy fails. For the treatment of intubation, there is still a lack of large-scale clinical trials to systematically explore its efficacy. The gradual increase in the clinical application of nHFOV has also enriched its use in the treatment of other diseases

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80, males and females;
2. Stage III and IV COPD and PaCO2≥50mmHg;
3. Similar with non-invasive ventilation;
4. Willing to participate in the study;
5. Able to provide informed consent.

Exclusion Criteria:

1. Bronchiectasis; post-tuberculosis sequelae; rib cage deformities; neuromuscular disorders; and bronchial carcinoma.
2. Intolerant with NIV

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Partial pressure of carbon dioxide in peripheral blood | within 50 minutes after intervention
  After the peripheral blood was arterialized for 10 minutes, 100 ul of the patient's finger peripheral blood was taken to measure the partial pressure of carbon dioxide in the peripheral blood.

SECONDARY OUTCOMES:
Asynchrony index | within 50 minutes after intervention
  Asynchrony index is defined as the number of asynchrony events divided by the total respiratory rate computed as the sum of the number of ventilator cycles (triggered or not) and of wasted efforts: asynchrony Index (expressed in percentage) = number of asynchrony events/total respiratory rate (ventilator cycles +wasted efforts) × 100